CLINICAL TRIAL: NCT01177995
Title: Fostering an AIDS Research and Training Center Infrastructure in Russia (Labor Migrant HIV Prevention Trial)
Brief Title: Russian Labor Migrant HIV Prevention Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yuri A. Amirkhanian, PhD, Associate Professor of Psychiatry and Behavioral Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R24MH082471 (NIH); R24MH082471 (NIH); PRO9948 (Other: Medical College of Wisconsin)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Social Network (Experimental): Leaders of labor migrant social networks will be trained to disseminate HIV prevention messages to the members of their social networks. The training will sequentially target ways to increase network members' HIV-related knowledge and norms, attitudes, intentions, and confidence in how to avoid risk. Leaders will be encouraged to have these discussions with network members between and after training sessions.
  Interventions: Behavioral: Social Network Intervention

INTERVENTIONS:
Behavioral: Social Network Intervention — Social network leaders will communicate HIV prevention messages to members of their social networks.

SUMMARY:
This study is a randomized outcome trial of a social network HIV prevention intervention for at-risk labor migrants who have arrived in St. Petersburg, Russia, to seek work. Most come to St. Petersburg from Moldova, Tajikistan, Uzbekistan, Ukraine, and other poor post-Soviet republics. While living in Russia, labor migrants are also living in a city and country with high HIV prevalence. Many labor migrants have limited awareness of AIDS, and most are living in a location far from their spouses, family members, and others. For that reason, labor migrants are vulnerable to risk behavior for contracting HIV.

This study hypothesizes that members of labor migrant social networks whose network leaders are trained to deliver HIV prevention messages will exhibit greater reductions in sexual risk behavior (unprotected intercourse with nonspousal partners) from baseline to 3- and 12-month followup assessments than will members of social networks whose members receive standard, individual HIV risk reduction counseling alone.

ELIGIBILITY:
Inclusion Criteria:

* being a labor migrant intending to temporarily work and reside in St. Petersburg, Russia, or being named as a member of the social network of a labor migrant;
* being at least 16 years old (the age at which persons can be legal labor migrants and are also legally considered to be able to provide informed consent);
* being able to complete written consent forms and questionnaire measures in Russian, Moldovan, Tajik, or Uzbek language
* providing written informed consent

Exclusion Criteria:

* being younger than age 16;
* not being able to complete written materials in the Russian, Moldovan, Tajik, or Uzbek language;
* planning to reside in St. Petersburg, Russia, for less than four months;
* having a severe mental or developmental disorder apparent by mental status during the study or consent explanation that, in the opinion of a trained interviewer, would preclude ability to understand informed consent or complete study measures

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Unprotected sexual intercourse events with a nonspousal partner | up to 12 months post intervention

SECONDARY OUTCOMES:
AIDS-related knowledge, attitudes, intentions, perceived norms, and self-efficacy | up to 12 months post intervention
  Factors reflecting HIV risk
Substance use related to sexual behavior | up to 12 months post intervention
  use of alcohol or other drugs in relation to sexual behavior

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A. Amirkhanian, PhD, Principal Investigator — Medical College of Wisconsin; Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin